CLINICAL TRIAL: NCT04881383
Title: The Development and Validation of a DM and Pre-DM Risk Prediction Function for Case Finding in Primary Care in Hong Kong
Brief Title: Development and Validation of DM and Pre-DM Risk Prediction Model
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Cindy L.K. Lam, Danny D. B. Ho Professor in Family Medicine and Head of Department, The University of Hong Kong
Other Study IDs: UW19-831
Record Dates: First submitted 2021-05-04; First posted 2021-05-11 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus; Pre Diabetes
Keywords: Risk prediction model; Early detection; Non-laboratory based
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients from Primary Care Clinics: Participating Chinese adults aged 18-84 from Primary Care clinics to validate the risk prediction function. Each subject will complete an assessment on the relevant risk factors and have a blood test on OGTT and HbA1c on recruitment and at 12 months.
  Interventions: Diagnostic Test: OGTT and HbA1c

INTERVENTIONS:
Diagnostic Test: OGTT and HbA1c — An investigation form will be given to the patient to attend an approved private laboratory for blood pressure, weight, height, waist and hip circumferences, and a blood test on OGTT, HbA1c, complete blood count (CBC) and lipid profile within three months

SUMMARY:
Many DM and pre-DM remain undiagnosed. The aim is to develop and validate a risk prediction function to detect DM and pre-DM in Chinese adults aged 18-84 in primary care (PC). The objectives are to:

1. Develop a risk prediction function using non-laboratory parameters to predict DM and pre-DM from the data of the HK Population Health Survey 2014/2015
2. Develop a risk scoring algorithm and determine the cut-off score
3. Validate the risk prediction function and determine its sensitivity in predicting DM and pre-DM in PC

Hypothesis to be tested:

The prediction function developed from the Population Health Survey (PHS) 2014/2015 is valid and sensitive in PC.

Design and subjects:

We will develop a risk prediction function for DM and pre-DM using data of 1,857 subjects from the PHS 2014/2015. We will recruit 1014 Chinese adults aged 18-84 from PC clinics to validate the risk prediction function. Each subject will complete an assessment on the relevant risk factors and have a blood test on OGTT and HbA1c on recruitment and at 12 months.

Main outcome measures:

The area under the Receiver operating characteristic (ROC) curve, sensitivity and specificity of the prediction function.

Data analysis and expected results:

Machine learning and Logistic regressions will be used to develop the best model. ROC curve will be used to determine the cut-off score. Sensitivity and specificity will be determined by descriptive statistics. A new HK Chinese general population specific risk prediction function will enable early case finding and intervention to prevent DM and DM complications in PC.

DETAILED DESCRIPTION:
Diabetes Mellitus (DM) is the second most common chronic non-communicable disease (NCD) and a major public health issue. In 2017, it was estimated that 451 million adults worldwide had DM, a number that is anticipated to rise to 693 million by 2045. In terms of economic burden, it was estimated that the global cost of DM in 2015 was 1·31 trillion US dollars, which accounted for 1.8% of global gross domestic product. In China, the prevalence of DM has increased rapidly, from less than 1% in 1980 to 10.9% in 2013, with approximately 109.6 million Chinese adults (25.8% of all cases worldwide) currently living with the condition. Among the Chinese population, Hong Kong has one of the highest prevalence of DM. The Population Health Survey (PHS) 2014/2015 conducted by Department of Health found a prevalence of 8.4% of DM among persons aged 15-84 in Hong Kong, more than half (4.5%) of which were previously unknown. Data (unpublished) from the Population Health Survey 2014/2015 showed a further 9.5% of persons aged 15-84 had hyperglycaemia (pre-diabetes) but were unaware of the problem before the survey DM can result in severe complications, which lead to disabling morbidity and premature mortality. A number of randomised controlled trials (RCTs) have found that lifestyle interventions (e.g., diet, exercise) and pharmacological treatments are effective in preventing DM and its complications. However, it has been reported that 224 million adults (49.7% of all cases) world-wide are unaware that they have the condition, similar to the finding of the Hong Kong PHS 2014/2015. DM can be present for 9-12 years prior to a diagnosis and is often only detected when patients present with complications. Hence, there is an urgent need for earlier detection of DM so that appropriate interventions can be provided to prevent and/or delay progression to complications. It would be even more effective if individuals could be identified at the pre-diabetes (pre-DM) stage when there may still be an opportunity to revert to normoglycaemia by life-style modifications. While DM satisfies all Wilson and Jungner's (1968) criteria of screening studies have shown that general population screening is not effective and the current recommendation is case finding targeting at high-risk individuals. The Hong Kong Reference Framework for Diabetes Care for Adults in Primary Care Settings recommends periodic screening for DM among persons aged >=45 years old or having DM risk factors. The recommended methods for screening include 75-g oral glucose tolerance tests (OGTT), fasting plasma glucose (FPG) tests or HbA1c tests. Indeed, a cost-effectiveness analysis reported that screening for DM and prediabetes was cost-saving among patients identified as being at high risk (e.g., body mass index (BMI) > 35 kg/m(2), systolic blood pressure ≥ 130mmHg or > 55 years of age) when compared with no screening. In order to identify high risk individuals more accurately, multivariate risk prediction models have been developed and incorporated into DM prevention programs in a number of Western countries. Such models have included sociodemographic factors (e.g., age, sex), clinical factors (e.g., family history of DM, gestational DM) or biomarkers (e.g., BMI, blood pressure). However, the majority of these models were developed primarily in Caucasian populations and have not performed as well among Chinese populations. For example, the Prospective Cardiovascular Münster, Cambridge, San Antonia and Framingham models were found to have inferior discrimination in a cohort of Chinese people. This can be due to ethnic differences as well as lifestyle and socioeconomic factors, calling for the need of population-specific risk prediction models. Since 2009, a number of risk prediction models and scoring algorithms have been developed specifically for Chinese populations, mostly from Mainland China, only two of which were developed and validated on Hong Kong Chinese people. The first used simple self-reported factors and laboratory measurements to develop a scoring algorithm. However, the generalisability of the model to primary care patients may be limited as 70% of the subjects of the development and validation samples had known risk factors for DM. The second risk prediction model for Hong Kong Chinese was previously developed by members of the investigators' team with data from 3,357 asymptomatic non-diabetic professional drivers. Non-laboratory risk factors included age, BMI, family history of DM, regular physical activity (PA), and high blood pressure. Triglyceride was added to the laboratory-based algorithm. The application of this risk predication model is limited because the sample was predominately male (92.7%) professional drivers and the accuracy was modest. It is noted that the majority of factors included in previous models are non-modifiable (e.g., family history of DM, gestational DM, age), and there is a call for future research to incorporate more lifestyle factors in order to improve the predictive validity and impact of risk prediction models. Lifestyle factors that may be associated with DM and pre-DM include physical activity (PA) level, dietary factors (e.g., fibre, sugar or fat intake), alcohol consumption, smoking and sleep. This proposed study aims to develop a new DM and pre-DM risk prediction model specific for the Hong Kong general Chinese population that incorporates traditional and modifiable life style factors. The investigators will apply the novel method of machine learning as well as the traditional logistic regression in model development to improve predictive power. The investigators hope the results will enable the implementation of effective case finding of DM and pre-DM in primary care, and prevent mortality and morbidity from this common but silent NCD for the people in Hong Kong.

ELIGIBILITY:
(Development Study)

Inclusion criteria:

* PHS 2014/2015 participants
* Completed the health examination including physical measurements (body height, weight, BMI, waist and hip circumference) and blood tests (fasting plasma glucose, HbA1c and lipid profile) during PHS 2014/2015
* aged 18-84 years

Exclusion criteria:

* Doctor-diagnosed DM
* Doctor-diagnosed high blood glucose
* Doctor-diagnosed cardiovascular disease (coronary heart disease, stroke)
* Doctor-diagnosed cancer
* Doctor-diagnosed chronic kidney disease
* Doctor-diagnosed anaemia

(Validation study)

Inclusion Criteria:

* Chinese
* aged 18-84 years
* Can communicate in Chinese
* Consent to participate in the study

Exclusion Criteria:

* Doctor-diagnosed DM
* Doctor-diagnosed high blood glucose
* Doctor-diagnosed cardiovascular disease (coronary heart disease, stroke)
* Doctor-diagnosed cancer
* Doctor-diagnosed chronic kidney disease
* Doctor-diagnosed anaemia
* Inability to complete the survey or blood test because of sickness or cognitive impairment
* Do not give consent to the study

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese adults aged 18-84 attending Primary Clinics clinics with no previous history of DM, CVD, cancer, CKD and anaemia
Sampling Method: Non-Probability Sample
Enrollment: 1014 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
The sensitivity of the risk prediction function in detecting DM and pre-DM in primary care | 12 months
  To validate the risk prediction functions, each of the models developed by logistic regressions or machine learning will be applied to the prospective data collected from subjects recruited from the participating primary care clinics. Overall sensitivity will be assessed by applying the risk threshold score to the validation data and a ROC curve of predicted risk against observed events (DM and pre-DM).

SECONDARY OUTCOMES:
Area under curve (AUC) of the risk prediction function in detecting DM and pre-DM in primary care | 12 months
  To validate the risk prediction functions, each of the models developed by logistic regressions or machine learning will be applied to the prospective data collected from subjects recruited from the participating primary care clinics. A ROC curve of predicted risk against observed events (DM and pre-DM) will be used to calculate the area under the curve (AUC) for assessing overall prediction accuracy.
Specificity of the risk prediction function in detecting DM and pre-DM in primary care | 12 months
  To validate the risk prediction functions, each of the models developed by logistic regressions or machine learning will be applied to the prospective data collected from subjects recruited from the participating primary care clinics. Overall specificity will be assessed by applying the risk threshold score to the validation data and a ROC curve of predicted risk against observed events (DM and pre-DM).
Positive predictive value (PPV) of the risk prediction function in detecting DM and pre-DM in primary care | 12 months
  To validate the risk prediction functions, each of the models developed by logistic regressions or machine learning will be applied to the prospective data collected from subjects recruited from the participating primary care clinics. Positive predictive value (PPV) will be assessed by applying the risk threshold score to the validation data and a ROC curve of predicted risk against observed events (DM and pre-DM).
Negative predictive value (NPV) of the risk prediction function in detecting DM and pre-DM in primary care | 12 months
  To validate the risk prediction functions, each of the models developed by logistic regressions or machine learning will be applied to the prospective data collected from subjects recruited from the participating primary care clinics. Negative predictive value (NPV) will be assessed by applying the risk threshold score to the validation data and a ROC curve of predicted risk against observed events (DM and pre-DM).

CONTACTS AND LOCATIONS:
Overall Officials: Cindy LK Lam, MD, Principal Investigator — Department of Family Medicine and Primary Care, University of Hong Kong
Locations (1):
- Department of Family Medicine & Primary Care, LKS Faculty of Medicine, University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Dong W, Cheng WHG, Tse ETY, Mi Y, Wong CKH, Tang EHM, Yu EYT, Chin WY, Bedford LE, Ko WWK, Chao DVK, Tan KCB, Lam CLK. Development and validation of a diabetes mellitus and prediabetes risk prediction function for case finding in primary care in Hong Kong: a cross-sectional study and a prospective study protocol paper. BMJ Open. 2022 May 24;12(5):e059430. doi: 10.1136/bmjopen-2021-059430. PMID 35613775